CLINICAL TRIAL: NCT03604744
Title: Direct Comparison of Altered States of Consciousness Induced by LSD and Psilocybin in a Random-order Placebo-controlled Cross-over Study in Healthy Subjects
Brief Title: Direct Comparison of Altered States of Consciousness Induced by LSD and Psilocybin
Acronym: LSD-psilo
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BASEC 2018-00985
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide; Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LSD-100, LSD-200, Psilocybin-15, Psilocybin-30, Placebo (Experimental): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Psilocybin
- LSD-200, Psilocybin-15, Psilocybin-30, Placebo, LSD-100 (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Psilocybin
- Psilocybin-15, Psilocybin-30, Placebo, LSD-100, LSD-200 (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Psilocybin
- Psilocybin-30, Placebo, LSD-100, LSD-200, Psilocybin-15 (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Psilocybin
- Placebo, LSD-100, LSD-200, Psilocybin-15, Psilocybin-30 (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Psilocybin

INTERVENTIONS:
Drug: LSD — LSD 0.1 mg per os, single dose
Drug: LSD — LSD 0.2 mg per os, single dose
Drug: Psilocybin — Psilocybin 15 mg per os, single dose
Drug: Psilocybin — Psilocybin 30 mg per os, single dose

SUMMARY:
LSD (lysergic acid diethylamide) and psilocybin (the active substance in "magic mushrooms") are widely used for recreational purposes. Both substances are also increasingly used in psychiatric and psychological research to induce and investigate alterations in waking consciousness and associated brain functions (functional brain imaging, "model psychosis") . However, it has never been studied whether there are differences in the alterations in mind produced by these two substances. Both LSD and psilocybin are thought to induce hallucinations primarily via stimulation of the 5-HT2A receptor. However, there are differences in the receptor activation profiles between the two substances that may also induce different subjective effects. LSD potently stimulates the 5-HT2A receptor but also 5-HT2B/C, 5-HT1 and D1-3 receptors . Psilocin (the active metabolite of the prodrug psilocybin) also stimulates the 5-HT2A receptor but additionally inhibits the 5-HT transporter. In contrast to LSD, psilocybin has no affinity for D2 receptors. Both substances are used in neuroscience as pharmacological tools. However, there are no modern studies comparing these two substances directly within the same clinical study and research subjects and using validated psychometric tools. Therefore, the investigators will compare the acute effects of LSD, psilocybin and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years.
2. Understanding of the German language.
3. Understanding the procedures and the risks that are associated with the study.
4. Participants must be willing to adhere to the protocol and sign the consent form.
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study.
6. Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
7. Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration.
8. Women of childbearing potential must have a negative pregnancy test at the beginning of the study. Pregnancy tests are repeated before each study session.
9. Women of childbearing potential must be willing to use double-barrier birth control
10. Body mass index 18-29 kg/m2.

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder in first-degree relatives
4. Illicit substance use (with the exception of cannabis) more than 10 times or any time within the previous two months.
5. Pregnant or nursing women.
6. Participation in another clinical trial (currently or within the last 30 days)
7. Use of medications that may interfere with the effects of the study medications (any psychiatric medications)
8. Tobacco smoking (>10 cigarettes/day)
9. Consumption of alcoholic drinks (>10/week)
10. Bodyweight < 50 kg

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Altered states of consciousness | 18 Months
  total 5D-ASC score (5-Dimensional Altered States of Consciousness Rating Scale)

SECONDARY OUTCOMES:
Subjective effects assessed by VAS | 18 Months
  VAS (Visual analog scale)
Subjective effects assessed by AMRS scales | 18 Months
  AMRS scales (Adjective mood Rating scale)
Psychotomimetic effects | 18 Months
  ESI (Eppendorf Schizophrenia Inventory)
Mystical-type experiences assessed by SCQ | 18 Months
  SCQ (States of consciousness questionnaire)
Mystical-type experiences assessed by MS scales | 18 Months
  MS scales (Mysticism scale)
Effects on emotion processing | 18 Months
  FERT (Face Emotion Recognition Task)
Autonomic effects assessed by heart rate | 18 Months
  Heart rate
Autonomic effects assessed by blood pressure | 18 Months
  Blood pressure (diastolic and systolic)
Autonomic effects assessed by body temperature | 18 Months
  Body temperature

OTHER OUTCOMES:
Plasma levels of LSD and psilocin | 18 Months
  assessment of plasma levels of LSD and psilocin

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holze F, Becker AM, Kolaczynska KE, Duthaler U, Liechti ME. Pharmacokinetics and Pharmacodynamics of Oral Psilocybin Administration in Healthy Participants. Clin Pharmacol Ther. 2023 Apr;113(4):822-831. doi: 10.1002/cpt.2821. Epub 2022 Dec 31. PMID 36507738
- [Derived] Holze F, Ley L, Muller F, Becker AM, Straumann I, Vizeli P, Kuehne SS, Roder MA, Duthaler U, Kolaczynska KE, Varghese N, Eckert A, Liechti ME. Direct comparison of the acute effects of lysergic acid diethylamide and psilocybin in a double-blind placebo-controlled study in healthy subjects. Neuropsychopharmacology. 2022 May;47(6):1180-1187. doi: 10.1038/s41386-022-01297-2. Epub 2022 Feb 25. PMID 35217796